CLINICAL TRIAL: NCT01336686
Title: A Phase 2 Randomized Double-Blind Placebo-Controlled Study to Evaluate the Safety and Efficacy of MBX-102 in the Treatment of Hyperuricemia in Patients With Gout
Brief Title: Safety and Efficacy Study of MBX-102 in Treatment of Hyperuricemia in Patients With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M102-21122
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Hyperuricemia; Gout
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — arhalofenate; Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arhalofenate 400 mg (Experimental)
  Interventions: Drug: Arhalofenate; Drug: Colchicine
- Arhalofenate 600 mg (Experimental)
  Interventions: Drug: Arhalofenate; Drug: Colchicine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo comparator; Drug: Colchicine

INTERVENTIONS:
Drug: Arhalofenate — Arhalofenate 400 mg once daily for 4 weeks
  Other Names: MBX-102
  Arms: Arhalofenate 400 mg
Drug: Arhalofenate — Arhalofenate 600 mg once daily for 4 weeks
  Other Names: MBX-102
  Arms: Arhalofenate 600 mg
Drug: Placebo comparator — Matching placebo once daily for 4 weeks
  Arms: Placebo
Drug: Colchicine — 0.6 mg colchicine daily for flare prophylaxis

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of MBX-102 compared to placebo when given orally once daily for 4 weeks for the treatment of hyperuricemia in patients with gout.

ELIGIBILITY:
Inclusion Criteria:

* Read and sign the informed consent after the elements of consent have been fully explained and all questions have been addressed, prior to any study procedures.
* Known gout patient (per criteria of the American Rheumatism Association for the classification of the acute arthritis of primary gout in Appendix 3)

  * the sUA must be ≥ 8.0 mg/dL and ≤12 mg/dL
  * if on ULT, the patients must agree to temporarily discontinue their existing ULT and the sUA must be ≥ 8.0 mg/dL and ≤12 mg/dL after wash-out at Week -1
* Male or female, 18-75 years of age at Screening Visit
* All female patients must be surgically sterile or post-menopausal (at least 45 years of age with no history of menses for at least 2 years; or any age with no history of menses for at least 6 months and serum FSH ≥ 40 mIU/mL) or have a partner who has undergone vasectomy or must agree to use two medically accepted methods of contraception including a barrier method (see the list in Appendix 4) for the entire duration of the study unless reporting complete sexual abstinence.
* Female patients must not be pregnant or lactating
* Male patients with a female partner of child-bearing potential must agree to use condom or the partner must use a medically acceptable method of contraception for the entire duration of the study.
* Patients must have an estimated CrCl ≥ 60 mL/min as calculated by the Cockcroft-Gault method
* Serum creatinine value must be ≤ 1.1 mg/dL in females and ≤ 1.3 mg/dL in males
* Patients must have liver function tests ≤ 1.5X ULN for AST, ALT and T-bilirubin, ≤ 2X ULN for ALP, ≤ 3X ULN for GGT; and ≤ 3X ULN for CK
* All other clinical laboratory parameters must be within normal limits or considered not clinically significant for participation in this study
* Electrocardiogram (ECG) must be normal, or if abnormal, considered not clinically significant for participation in this study
* Patients must have a systolic blood pressure ≤ 160 mm Hg and a diastolic blood pressure ≤ 90 mm Hg; known hypertensive patients controlled with medication other than thiazide diuretics (BP reading as above) may be included

Exclusion Criteria:

* Known or suspected secondary hyperuricemia (e.g. due to myeloproliferative disorder, or organ transplant).
* Known patient with xanthinuria
* History of documented or suspected kidney stones
* Over producers of uric acid as evidenced by 24-hour urinary uric acid > 800 mg (on normal unrestricted diet)
* Known infection with the human immunodeficiency virus (HIV) or history of viral hepatitis type B or C
* History of illicit drug or alcohol abuse within last 1 year
* History of significant pulmonary disease, upper GI bleeding, documented peptic ulcer disease (unless known H. pylori infection treated successfully without recurrence), or nephrotic syndrome within last 3 years
* All patients must not have had a stroke, TIA, acute myocardial infarction, congestive heart failure (NYHA Class II-IV), angina pectoris, coronary intervention procedure (including but not limited to angioplasty, stent placement, coronary revascularization), lower extremity bypass procedure, systemic or intracoronary fibrinolytic therapy within last 5 years
* Malignancy within the last 5 years (except resected basal cell carcinoma)
* Body mass index (BMI) > 42 kg/m2
* Current or expected requirement for anticoagulant therapy (except for ≤ 325 mg/day aspirin and/or Plavix® 75 mg/day)
* Rheumatoid arthritis or other autoimmune disease requiring ongoing treatment
* Current or expected treatment with potent CYP3A4 inhibitors (See in Appendix 6), ranolazine, digoxin, cyclosporine, cyclophosphamide and other cytotoxic agents, sulphonylurea, thiazolidinedione, diuretic, atypical antipsychotic agents, and phenytoin
* Chronic treatment with non-steroidal anti-inflammatory drugs (NSAIDs use to treat acute flares are permitted)
* Current or expected treatment with systemic corticosteroids (except topical, ophthalmic, intra-articular, or inhaled at a dose < 1600 μg/day) other than to treat acute flares
* Known hypersensitivity to colchicine
* Treatment with any other investigational therapy within the 30 days prior to the Screening Visit, or patients who received at least one dose of blinded study drug while enrolled in any previous MBX-102 trial
* Any other condition that compromises the ability of the patient to provide informed consent or to comply with the objectives and procedures of this protocol, as judged by the investigator and/or medical monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Serum uric acid | Baseline and end of treatment phase (4 wks)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Tucson, Arizona
  - Los Angeles, California
  - Boca Raton, Florida
  - Jupiter, Florida
  - Tampa, Florida
  - Honolulu, Hawaii
  - Wheaton, Maryland
  - St Louis, Missouri
  - New York, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - West Jordan, Utah